CLINICAL TRIAL: NCT02581358
Title: Use of the Scolioscan for Quantitative Evaluation of Spinal Deformity - A Validity Study on Patients With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Assistant Professor (Clinical), Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PhaseIII_V.3
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Scoliosis
Keywords: scoliosis; spinal deformity; Cobb angle; assessment; ultrasound
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scolioscan (Ultrasound imaging system) (Experimental): This diagnostic study is a single arm study with all participants receiving investigation with the Scolioscan (a diagnostic ultrasound machine) for quantitative assessment of spinal deformity
  Interventions: Other: Scolioscan (Ultrasound imaging system)

INTERVENTIONS:
Other: Scolioscan (Ultrasound imaging system) — To assess the scoliotic patient, a 3D ultrasound imaging system (the Scolioscan) was developed. The system composes of an ultrasound scanner with a linear probe, a frame structure, an electromagnetic spatial sensing device and a dedicated PC program for imaging and data collection, processing, visualization, analysis, and assessment. The spatial sensor was attached to the ultrasound probe for spatial information collection and calibration. The Scolioscan will generate ultrasound images of the spine for quantitative assessment of the curve deformity in terms of Cobb angles.

SUMMARY:
The purpose of the study is to investigate the validity of Scolioscan for quantitative assessment of curve severity in scoliosis using x-ray radiographs as the gold standard.

DETAILED DESCRIPTION:
Scoliosis is a three dimensional spinal deformity, in both the coronal plane, sagittal and transverse planes. Quantitative assessment of curve severity in scoliosis is important for patient management. At present, Cobb angle measurement in the frontal plane using standing postero-anterior X-ray radiograph is the gold standard for scoliosis evaluation. Taking x-ray involves irradiation and is not without risk especially over repeated exposures for follow-up visits. With advancement of ultrasound technology which is radiation-free and noted to be useful as a tool for musculoskeletal imaging, an ultrasound system designed for evaluation of spinal deformity called Scolioscan has been developed. It comprises of a freehand 3D ultrasound imaging system with an enhanced frame structure for supporting the patient to maintain the posture during scanning and a software for measuring curve deformity in terms of Cobb angles. Previous studies on validity of ultrasound assessment for back deformity involved a pilot group of subjects. Based on these promising pilot results, we plan to carry out a formal study to investigate the validity of Scolioscan for quantitative assessment of curve severity in scoliosis using x-ray radiograph as the gold standard for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis patients between 8-40 years old
* Patients with body mass index (BMI) <23 kg/m2
* Patients with standing height between 1 m - 2 m

Exclusion Criteria:

* Pregnant women or women after pregnancy before return of the menstrual period.
* Subjects with skin disease such as skin cancer, psoriasis or a history of skin disease
* Subjects with fracture or wound that affect application of the probe of Scolioscan during scanning
* Subjects with Ferromagnetic implants
* Subjects with pacemakers, implanted pain modulators, implanted insulin delivery systems, cochlear implant, and any defibrillator
* Subjects with surgery done for the spine
* Subjects with winged scapula or other irregularity of back contour that precludes satisfactory skin contact of the machine probe during the scanning procedure
* Subjects who cannot stand steadily on the device during the examination
* Subjects with allergy to aqueous gel used for ultrasound scanning

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 952 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cobb angle | Baseline
  Curve deformity measurement in terms of Cobb angles assessed by Scolioscan will be correlated with those assessed with conventional x-ray radiographs. The correlation will be compared between:
  1. mild and severe curves
  2. thoracic and lumbar curves
  3. low BMI and high BMI subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ping Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, Hong Kong, Hong Kong, China